CLINICAL TRIAL: NCT01843842
Title: Multicentre Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Safety and Clinical Efficacy of Ergoferon in Liquid Dosage Form in Treatment of Acute Upper Respiratory Tract Infections in Children
Brief Title: Clinical Trial of Safety and Clinical Efficacy of Ergoferon in Liquid Dosage Form in Treatment of Acute Upper Respiratory Tract Infections in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-ER-007
Record Dates: First submitted 2013-04-26; First posted 2013-05-01 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Acute Upper Respiratory Tract Infections
MeSH Terms: interventions — ergoferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergoferon (5 ml 3 times a day) (Experimental)
  Interventions: Drug: Ergoferon
- Placebo (5 ml 3 times a day) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergoferon — Safety and Efficiency of liquid dosage form
  Arms: Ergoferon (5 ml 3 times a day)
Drug: Placebo — Safety and Efficiency of liquid dosage form
  Arms: Placebo (5 ml 3 times a day)

SUMMARY:
The purpose of this study is:

* to assess safety of the liquid dosage form of Ergoferon for treatment of acute upper respiratory tract infections in children;
* to assess clinical efficacy of the liquid dosage form of Ergoferon for treatment acute upper respiratory tract infections in children.

DETAILED DESCRIPTION:
The overall duration of a patient's participation in the trial is 6 days (screening/randomization, therapy onset - day 1; study therapy period - 5 days; follow-up period-1 day).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged over 3 years and under 18 years.
2. Patients who consulted a doctor within 24 hours after the onset of acute respiratory infection (body temperature no less than 38.0°C when visiting a doctor + intensity of symptoms ≥ 4 scores (presence of at least 1 general symptom ≥ 2 scores and 1 nasal/ throat/ chest symptom ≥ 2 scores or greater number of symptoms with the intensity≥1 score) during seasonal morbidity.
3. The possibility to start therapy within 24 hours after the onset of the first symptoms of acute respiratory infection.
4. Usage of contraceptive methods by sexually active teenagers of both sexes during the trial and within 30 days after ending of the participation in the trial.
5. Availability of information sheet (Informed Consent form) for parents/adopters of patient for participation in the clinical trial, Version 2.1 or Version 2.2, signed by one parent/adopter of patient. For patients over 14 years - availability of information sheet (Informed Consent form) for participation in the clinical trial, Version 2.1 or Version 2.2, signed by a patient and one parent/adopter of patient.

Exclusion Criteria:

1. Suspected bacterial infection or presence of a severe disease requiring use of antibacterial drugs (including sulfanilamides).
2. Suspected initial manifestations of diseases that have symptoms similar to acute respiratory infection (other infectious diseases, influenza-like syndrome at the onset of systemic connective tissue disorders, oncohematology and other pathology).
3. Medical history of primary and secondary immune deficiency: a) lymphoid system immunodeficiency (T-cell and /or B-cell immunity chain, immunodeficiency with predominant antibody deficiency); b) phagocyte deficiency; c) complement factors deficiency; d ) combined immunodeficiency including AIDS induced by HIV infection; toxic, autoimmune, infectious, radial panleukopenia syndrome; general lymphocytopenia syndrome; syndrome of lymphocyte polyclonal activation; postsplenectomia syndrome; congenital asplenia; syndrome of immune complexes pathology associated with infectious, allergic and autoimmune diseases.
4. Medical history of sarcoidosis.
5. Oncological diseases.
6. Exacebration or decompensation of chronic diseases affecting the patient's ability to participate in the clinical trial.
7. Medical history of polyvalent allergy.
8. Allergy/ intolerance to any of the components of medications used in the treatment.
9. Impaired glucose tolerance, diabetes mellitus.
10. Hereditary fructose intolerance (as the study drug contains maltitol).
11. Intake of medicines listed in the section "Prohibited concomitant treatment" for 1 month prior to the inclusion in the trial.
12. Pregnancy, unwillingness of sexually active female patients to use of contraceptive methods during the study.
13. Drug addiction, alcohol usage in the amount 2 units of alcohol per day on the part of patient's parents/adopters.
14. Mental disorders of patient or of patient's parents/adopters.
15. Patient's parents/ adopters, who from investigator's point of view, will fail to comply with the observation requirements of the trial or with the intake regimen of the investigated medicines.
16. Participation in other clinical trials in the course of 3 months prior to the inclusion in the trial.
17. Patient's parent/adopter is related to the research personnel of the investigative site, who are directly involved in the trial or are the immediate relative of the researcher. The immediate relatives includes husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
18. Patient's parent/adopter works for OOO "NPF "Materia Medica Holding" (i.e. is the company's employee, temporary contract worker or appointed official responsible for the carrying out the research) or the immediate relative.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 306 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - State Educational Institution of Higher Professional Education "Moscow State Medical Academy named after I.M. Sechenov", Moscow
  - State Budgetary Educational Institution of Higher Professional Education Novosibirsk State Medical University of Ministry of Health of Russian Federation, Novosibirsk
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №5", Perm
  - St. Peterburg State Health Care Institution "Child Health City Hospital №45 of the Nevsky Region", Saint Peterburg
  - State Budgetary Health Care Institution "Сity Child Health Polyclinic №44", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic №44", Saint Petersburg
  - State Budgetary Educational Institution of Higher Professional Education "St. Petersburg State Pediatric Medical Academy" of Ministry of Health of Russian Federation, Saint Petersburg
  - Limited Liability Company "Alliance Biomedical-Russian group", Saint Petersburg
  - State Health Care Institution "Child Health City Hospital №22", Saint Petersburg
  - State Budgetary Educational Institution of Higher Professional Education " Yaroslavl State Medical Academy" of Ministry of Health, Yaroslavl
  - Municipal Institution "Child Health City Hospital №11", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon in Liquid Dosage Form: Children aged 3 to 18 years were on the treatment regimen with Ergoferon in Liquid Dosage Form for 5 days. 1 dosing spoon (5 ml) per 1 intake: on day 1 of the treatment 8 dosing spoons (1 dosing spoon every 30 minutes for the first 2 hours, then 1 dosing spoon 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 dosing spoon tablet 3 times a day.
- Placebo: Children aged 3 to 18 years were on the treatment regimen with Placebo for 5 days. 1 dosing spoon (5 ml) per 1 intake: on day 1 of the treatment 8 dosing spoons (1 dosing spoon every 30 minutes for the first 2 hours, then 1 dosing spoon 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 dosing spoon tablet 3 times a day.
Period: Overall Study
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Started | 154 | 152
Completed | 153 | 151
Not Completed | 1 | 1
Not completed — Do not meet inclusion criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ergoferon in Liquid Dosage Form; Placebo: 1 dosing spoon (5 ml) per 1 intake: on day 1 of the treatment 8 dosing spoons (1 dosing spoon every 30 minutes for the first 2 hours, then 1 dosing spoon 3 times a day with equal intervals starting on the same day. From day 2 to day 5 1 dosing spoon tablet 3 times a day
- Total: Total of all reporting groups
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo | Total
Number analyzed (Participants) | 154 | 152 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (4.1) | 10.2 (4.2) | 10.0 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 80 | 147
  Male | 87 | 72 | 159
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 154 | 152 | 306

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Recovery/Improvement in Health on Days 2, 3 and 4 of Observation (Based on Patient Diary Data)
Description: Based on the data mentioned in a patient's diary
Time Frame: On day 2, 3 and 4 of observation
Population: Per Protocol set
Measure: Number; unit: percentage of participants
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
percentage of participants
  Day 2 | 9 | 1
  Day 3 | 21 | 11
  Day 4 | 44 | 33
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Test type: Superiority; p = 0.016, Global Test Statistic; See O'Brien 1984, Pocock 1997

2. Secondary Outcome: Dynamics of Fever (Changes in Body Temperature on 2, 3, 4, 5 Days of Observation in Comparison With the Baseline)
Time Frame: baseline and days 2, 3, 4 and 5 of observation
Population: Per Protocol set. The morning temperature in 13 patients (7 in the Ergoferon group and 6 in the placebo group) was excluded from the analysis due to mistakes in diaries.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 138 | 142
°C
  Day 2, Morning | -0.96 (0.55) | -0.79 (0.53)
  Day 3, Morning | -1.49 (0.47) | -1.30 (0.50)
  Day 4, Morning | -1.77 (0.41) | -1.69 (0.44)
  Day 5, Morning | -1.90 (0.37) | -1.86 (0.38)
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

3. Secondary Outcome: Percentage of Patients With Normal Body Temperature (≤37.0ºС)
Description: Axillary temperature (morning and evening) decline to or below 37.0 ºС
Time Frame: On day 2, 3, 4, 5 of observation
Population: Per Protocol set.
Measure: Number; unit: percentage of participants
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
percentage of participants
  Day 2, Morning | 21 | 16
  Day 2, Evening | 29 | 22
  Day 3, Morning | 68 | 53
  Day 3, Evening | 59 | 51
  Day 4, Morning | 89 | 86
  Day 4, Evening | 81 | 78
  Day 5, Morning | 98 | 97
  Day 5, Evening | 94 | 95
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Test type: Superiority; p > 0.05, Fisher Exact

4. Secondary Outcome: Severity of Clinical Manifestations of Acute Respiratory Infection (ARI) by Total Symptom Score on Day 3 of Observation (Based on the Results of Pediatrician's Examination) and on Days 2, 3, 4 and 5 of Observation (Based on Patient Diary Data)
Description: The Total Symptom Score (TSS) was based on the severity of each of acute respiratory infection (ARI) symptom.
  The TSS includes 13 symptoms: Body temperature / fever, Non-specific ARI symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), Nasal/Throat/Chest symptoms (Runny nose, Nasal congestion, Sneezing, Sore throat, Hoarseness, Cough, Chest pain/Tightness of the chest).
  The severity of Non-specific and Nasal/Throat/Chest symptom was scored on a symptom severity scale (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms). The Fever was scored on a symptom severity scale 0 = no symptom (≤37,30С); 1 = mild symptom (37,4-38,00С); 2 = moderate symptom (38,1-39,00); 3 = severe symptom (≥39,10С).
  Minimum score=0; maximum score=39. The severity of ARI symptoms was recorded: 1) by the doctors on the case record form on Day 3; 2) by one of the patient's parents/adopter on a diary card twice a day (morning and evening) on Days 2-5.
Time Frame: on Days 2, 3, 4, 5 of Observation
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
Score
  Fever (Day 3, doctor's examination) | 0.3 (0.5) | 0.4 (0.6)
  Non-specific (Day 3, doctor's examination) | 1.7 (1.8) | 1.9 (1.8)
  Nasal/Throat/Chest (Day 3, doctor's examination) | 3.6 (2.2) | 3.7 (2.1)
  All symptoms (Day 3, doctor's examination) | 5.5 (3.7) | 6.0 (3.6)
  Fever (Day 2, patient diary data) | 0.8 (0.7) | 1.0 (0.8)
  Non-specific (Day 2, patient diary data) | 3.3 (3.0) | 4.1 (3.1)
  Nasal/Throat/Chest (Day 2, patient diary data) | 4.4 (2.8) | 5.0 (2.8)
  All symptoms (Day 2, patient diary data) | 9.4 (6.1) | 11.1 (6.3)
  Fever (Day 3, patient diary data) | 0.3 (0.5) | 0.5 (0.6)
  Non-specific (Day 3, patient diary data) | 1.7 (1.9) | 1.9 (1.8)
  Nasal/Throat/Chest (Day 3, patient diary data) | 3.3 (2.2) | 3.6 (2.1)
  All symptoms (Day 3, patient diary data) | 5.6 (4.2) | 6.4 (4.1)
  Fever (Day 4, patient diary data) | 0.1 (0.3) | 0.1 (0.4)
  Non-specific (Day 4, patient diary data) | 0.6 (1.1) | 0.8 (1.2)
  Nasal/Throat/Chest (Day 4, patient diary data) | 2.3 (2.0) | 2.3 (1.4)
  All symptoms (Day 4, patient diary data) | 3.1 (2.9) | 3.3 (2.5)
  Fever (Day 5, patient diary data) | 0.0 (0.2) | 0.0 (0.2)
  Non-specific (Day 5, patient diary data) | 0.2 (0.8) | 0.2 (0.6)
  Nasal/Throat/Chest (Day 5, patient diary data) | 1.3 (1.5) | 1.3 (1.2)
  All symptoms (Day 5, patient diary data) | 1.6 (2.0) | 1.6 (1.7)
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Fever (Day 3, doctor's examination); Test type: Superiority; p = 0.0283, Kruskal-Wallis — p-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Non-specific (Day 3, doctor's examination); Test type: Superiority; p = 0.3264, Kruskal-Wallis
Statistical Analysis 3: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Nasal/Throat/Chest (Day 3, doctor's examination); Test type: Superiority; p = 0.7060, Kruskal-Wallis
Statistical Analysis 4: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; All symptoms (Day 3, doctor's examination); Test type: Superiority; p = 0.25, Kruskal-Wallis
Statistical Analysis 5: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Severity of clinical manifestations of acute respiratory infection (ARI) by Total Symptom Score on Days 2, 3, 4 and 5 of Observation (Based on Patient Diary Data); Test type: Superiority; p = 0.244, ANCOVA

5. Secondary Outcome: Duration of Acute Respiratory Infection Symptoms (Fever, Non-specific Symptoms and Nasal/ Throat/ Chest Symptoms) Based on Patient Diary Data
Description: Acute respiratory infection (ARI) symptoms include 13 symptoms: Body temperature / fever, Non-specific ARI symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), Nasal/Throat/Chest symptoms (Runny nose, Nasal congestion, Sneezing, Sore throat, Hoarseness, Cough, Chest pain/Tightness of the chest).
  The ARI symptoms was recorded by one of the patient's parents/adopter on a diary card twice a day (morning and evening) on Days 1-5.
Time Frame: baseline and days 2, 3, 4 and 5 of observation
Population: Per Protocol set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
hours
  Fever | 26.7 (22.9) | 31.6 (23.9)
  Non-specific symptoms | 55.2 (31.0) | 60.8 (30.5)
  Nasal/ throat/ chest symptoms | 84.0 (33.2) | 88.9 (29.9)
  All symptoms | 86.0 (30.8) | 91.1 (27.9)
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Duration of fever based on Patient Diary Data; Test type: Superiority; p = 0.1158, Kruskal-Wallis
Statistical Analysis 2: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Duration of non-specific symptoms based on Patient Diary Data; Test type: Superiority; p = 0.5755, Kruskal-Wallis
Statistical Analysis 3: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Duration of nasal/ throat/ chest symptoms based on Patient Diary Data; Test type: Superiority; p = 0.4331, Kruskal-Wallis
Statistical Analysis 4: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Duration of all acute respiratory infection symptoms (fever, non-specific symptoms and nasal/ throat/ chest symptoms) based on Patient Diary Data; Test type: Superiority; p = 0.3560, Kruskal-Wallis

6. Secondary Outcome: Severity of the Disease Within 6 Days Was Assessed Using the "Area Under the Curve" for the Total Symptom Score (TSS)
Description: The Total Symptom Score (TSS) was based on the severity of each of acute respiratory infection (ARI) symptom.
  The TSS includes 13 symptoms: Body temperature / fever, Non-specific ARI symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), Nasal/Throat/Chest symptoms (Runny nose, Nasal congestion, Sneezing, Sore throat, Hoarseness, Cough, Chest pain/Tightness of the chest).
  The severity of Non-specific and Nasal/Throat/Chest symptom was scored on a symptom severity scale (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms). The Fever was scored on a symptom severity scale 0 = no symptom (≤37,30С); 1 = mild symptom (37,4-38,00С); 2 = moderate symptom (38,1-39,00); 3 = severe symptom (≥39,10С).
  Minimum score=0; maximum score=39. The severity of ARI symptoms was recorded: 1) by the doctors on the case record form on Days 1, 3, 6; 2) by one of the patient's parents/adopter on a diary card twice a day (morning and evening) on Days 1-5.
Time Frame: On days 1-6 of observation
Population: Per Protocol set.
Measure: Mean (Standard Deviation); unit: AUC score*day
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
AUC score*day
  Fever (Days 1, 3, 6 doctor's examination) | 1.3 (0.6) | 1.5 (0.7)
  Non-specific (Days 1, 3, 6 doctor's examination) | 4.9 (3.0) | 5.2 (2.6)
  Nasal/Throat/Chest (Days 1, 3, 6 doctor's examinat | 6.9 (3.6) | 7.2 (3.3)
  All symptoms (Days 1, 3, 6 doctor's examination) | 13.1 (5.7) | 13.9 (5.3)
  Fever (Days 1-5, patient diary data) | 2.1 (1.6) | 2.6 (1.7)
  Non-specific (Days 1-5, patient diary data) | 8.7 (6.7) | 10.1 (6.6)
  Nasal/Throat/Chest (Days 1-5, patient diary data) | 13.4 (8.0) | 14.4 (7.1)
  All symptoms (Days 1-5, patient diary data) | 26.3 (14.8) | 29.6 (14.1)
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Fever (Days 1, 3, 6 doctor's examination); Test type: Superiority; p = 0.0166, Kruskal-Wallis — p-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Non-specific (Days 1, 3, 6 doctor's examination); Test type: Superiority; p = 0.0820, Kruskal-Wallis
Statistical Analysis 3: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Nasal/Throat/Chest (Days 1, 3, 6 doctor's examination); Test type: Superiority; p = 0.7227, Kruskal-Wallis
Statistical Analysis 4: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; All symptoms (Days 1, 3, 6 doctor's examination); Test type: Superiority; p = 0.2645, Kruskal-Wallis
Statistical Analysis 5: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Fever (Days 1-5, patient diary data); Test type: Superiority; p = 0.0142, Kruskal-Wallis — p-value is not adjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Non-specific (Days 1-5, patient diary data); Test type: Superiority; p = 0.0145, Kruskal-Wallis — p-value is not adjusted for multiple comparisons
Statistical Analysis 7: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Nasal/Throat/Chest (Days 1-5, patient diary data); Test type: Superiority; p = 0.2963, Kruskal-Wallis
Statistical Analysis 8: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; All symptoms (Days 1-5, patient diary data); Test type: Superiority; p = 0.0364, Kruskal-Wallis — p-value is not adjusted for multiple comparisons

7. Secondary Outcome: Number of Intakes of Antipyretics if Indicated
Description: Based on data mentioned in a patient's diary
Time Frame: On day 1, 2, 3, 4 and 5 of the treatment
Population: Per Protocol set.
Measure: Mean (Standard Deviation); unit: Number of intakes
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
Number of intakes
  Day 1 | 0.84 (0.86) | 0.85 (0.78)
  Day 2 | 0.20 (0.57) | 0.30 (0.71)
  Day 3 | 0.08 (0.36) | 0.09 (0.40)
  Day 4 | 0.03 (0.26) | 0.03 (0.25)
  Day 5 | 0.01 (0.17) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Ergoferon in Liquid Dosage Form vs Placebo; Test type: Superiority; p = 0.40, ANCOVA

8. Secondary Outcome: Percentage of Patients With Exacerbation of the Disease Course
Description: The development of disease complications requiring antibiotics administration or hospitalization
Time Frame: On days 1-6 of observation
Population: Per Protocol set.
Measure: Number; unit: percentage of participants
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Number analyzed (Participants) | 145 | 148
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered from Day 1 to Day 6
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=306, Safety Population)
Arm/Group | Ergoferon in Liquid Dosage Form | Placebo
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/152
Other Adverse Events (participants affected / at risk) | 3/154 | 2/152
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ergoferon in Liquid Dosage Form (N=154) | Placebo (N=152)
Ear ache (Ear and labyrinth disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Disturbance of a night's sleep (Psychiatric disorders) | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other